CLINICAL TRIAL: NCT04242212
Title: A Prospective, Comparative Study of Clinical Outcomes Following Clinic-based Versus Self-use of Medication Abortion Using a Misoprostol-only Regimen
Brief Title: Study of Clinic-based vs. Self-use of a Misoprostol-only Regimen for Induced Abortion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ipas (Other)
Responsible Party: Sponsor
Other Study IDs: Ipas_NMAS
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Induced Abortion; First Trimester Abortion
Keywords: Medication abortion; Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinic-based: Women who get misoprostol from a clinic-based provider
  Interventions: Behavioral: Misoprostol sourced from clinics
- PMV-based: Women who get misoprostol from a patent medicine vendor
  Interventions: Behavioral: Misoprostol sourced from PMVs

INTERVENTIONS:
Behavioral: Misoprostol sourced from clinics — One cohort of women using misoprostol sourced from clinics
  Groups: Clinic-based
Behavioral: Misoprostol sourced from PMVs — One cohort of women using misoprostol sourced from PMVs
  Groups: PMV-based

SUMMARY:
The goal of the study is to determine whether important clinical outcomes differ among women who access a misoprostol-only medication abortion regimen from a patent medicine vendor when compared with those who access it from a clinic.

DETAILED DESCRIPTION:
Medication abortion with a misoprostol-only regimen within the first 10 weeks of pregnancy is safe and effective. Investigators aim to assess whether self-use of early (<9 weeks) medication abortion using a misoprostol-only regimen results in non-inferior rates of clinical outcomes when compared with clinic-based provision of medication abortion.

The investigators will prospectively recruit women who obtain misoprostol from patent medicine vendors and clinics. Follow-up will occur by telephone during three phone calls within 45 days of the first dose of misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Purchased a misoprostol-only abortion regimen at a PMV or from a clinic
* Be at least 15 years of age
* Have a known LMP of less than 9 weeks
* No contraindications to medical abortion
* Willing and able to give informed consent
* Have a mobile phone of which they are the independent user or be willing to be followed-up in person
* Willing to be contacted with questions about her abortion by telephone at 1-3, 10-29 and 30-45 days following initial contact.

Exclusion Criteria:

* Contraindications to misoprostol
* Age <15 or >49

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Nigerian women, age 15-49, living in the study geography, who are pregnant and seeking a misoprostol-only regimen for medication abortion, either from a patent medicine vendor or a healthcare clinic/facility.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-05-19 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Need for additional treatment to complete abortion | Final assessment at 45 days following misoprostol
  The primary outcome of the study will be the need for additional treatment to complete the abortion (either aspiration or repeated misoprostol >3 doses) following a woman taking the medication abortion pills.

SECONDARY OUTCOMES:
Serious complications/ morbidity | Final assessment at 45 days following misoprostol
  Number of participants who have a complication such as hemorrhage requiring a blood transfusion, hospitalization, serious infection and undiagnosed (at the time of misoprostol) ectopic pregnancy.

OTHER OUTCOMES:
Uptake of postabortion contraception | Final assessment at 45 days following misoprostol
  Women's reported use of contraception (yes or no and method type) following medication abortion.

CONTACTS AND LOCATIONS:
Locations (3):
- Nigeria (3):
  - Multiple facilities, Awka, Anambra
  - Multiple facilities, Abeokuta, Ogun State
  - Multiple facilities, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: No